CLINICAL TRIAL: NCT06497010
Title: An Open Label, Prospective, Exploratory Study to Assess the Safety and Efficacy of Individualized Neo-antigen mRNA Cancer Vaccine InnoPCV in Combination With PD-1 in Participants With Advanced Solid Tumor
Brief Title: An Exploratory Study of Individualized Neo-antigen mRNA Cancer Vaccine InnoPCV in Advanced Solid Tumor Treatment
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Collaborators: Innovac Therapeutics (Industry)
Responsible Party: Principal Investigator, Shengfa Su, Chief Physician, The Affiliated Hospital Of Guizhou Medical University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: InnoPCV-001
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Experimental): Part A (PD-1 Run-in):
  Participants will receive either tislelizumab (200 mg, IV Q3W) or sintilimab (200 mg, IV Q3W) for a lead-in period of one to three cycles.
  Part B( InnoPCV in Combination with PD-1)：
  Participants will commence up to nine cycles of combination therapy, consisting of InnoPCV (0.06 - 1 mg, intramuscularly, every three weeks) in conjunction with the anti-PD-1 antibody (200 mg, intravenous infusion, every three weeks).
  Part C (PD-1 maintenance treatment)
  Participants will continue with maintenance therapy using either tislelizumab (200 mg, IV Q3W) or sintilimab (200 mg, IV Q3W) until disease progression or unacceptable toxicity observed
  Interventions: Drug: Biological: PD-1; Drug: Biological: InnoPCV

INTERVENTIONS:
Drug: Biological: PD-1 — Intravenous (IV) infusion
Drug: Biological: InnoPCV — Intramuscular (IM) injection

SUMMARY:
This is an open-label, prospective, exploratory clinical study, which is divided into two phases: dose escalation phase (Phase Ia) and expansion phase (Phase Ib). After completing the dose-escalation phase (Stage Ia) (5-11 patients), the investigator will select the dose group (RP2D) based on safety, tolerability, and preliminary immune-related characteristics and efficacy data, and choose 2-3 advanced solid tumors to enter the expansion phase (Stage Ib).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, male or female.
* Histologically/cytologically or clinically confirmed advanced unresectable protocol-specified solid malignancies.
* Participants with Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Life expectation >= 12weeks.
* Participants must have a formalin-fixed paraffin-embedded (FFPE) tumor sample available (for example, from their prior surgery) that is suitable for the next-generation sequencing (NGS) required for this study.
* Adequate organ function.
* Participants must agree to use adequate contraception from the first dose of study medication through 180 days after the last dose of study medication (male and female participants of childbearing potential).

Exclusion Criteria:

* Not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the adverse events (except for alopecia, vitiligo, neurotoxicity, hypothyroidism hormone replacement therapy) caused by therapy administered within 4 weeks before the first dose of PD-1.
* Participants with a history of (non-study tumor) malignancy (except for skin squamous cell carcinoma and basal cell carcinoma, in situ cervical or breast carcinoma) within 3 years before the first dose of PD-1.
* Participation in a study of an investigational agent or using an investigational device within 30 days before the first dose of PD-1.
* Previously received any adoptive cell therapy (including but not limited to tumor-infiltrating lymphocyte TILs, chimeric antigen receptor T cells (CAR-T) and T cell receptor chimeric T cells (TCR-T)), therapeutic tumor vaccines, etc.
* Participants received chemotherapy, radiotherapy (palliative radiotherapy is allowed), and immune activator (including but not limited to IL-2) and other antitumor therapy within 21 days before the first dose; Participants received Chinese herbal medicine within 2 weeks before the first dose of PD-1.
* Major surgery (excluding diagnostic biopsy) or significant trauma had not been fully recovered within 28 days before the first dose of PD-1.
* Participants received live attenuated vaccine within 28 days before starting study treatment or planned to receive live attenuated vaccine during the study and within 60 days after ending the study drug treatment.
* Active autoimmune disease or a documented history of autoimmune disease or the syndrome that requires systemic steroids or immunosuppressive agents, except vitiligo or resolved childhood asthma/atopy.
* Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (HBV-DNA≥ 500IU/ml), or Hepatitis C virus (Hepatitis C Virus Ribonucleic Acid [HCV RNA] (qualitative) is detected).
* Previously identified hypersensitivity to components of the formulations used in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Baseline through 90 days after last InnoPCV dose

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Baseline through 90 days after last tislelizumab or sintilimab dose
Neoantigen-specific T cell Response rate | Baseline through 26 weeks after last InnoPCV dose
Objective Response Rate (ORR): Number of Participants with Tumor Response (Partial or Complete) | Baseline through disease progression by Response Evaluation Criteria of Solid Tumors Version 1.1 (RECIST 1.1), start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 2 years)
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR).
Duration of Response (DoR) | Baseline through disease progression by Response Evaluation Criteria of Solid Tumors Version 1.1 (RECIST 1.1), start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 2 years)
  DoR is defined as time from first tumor response (partial or complete) until either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Progression Free Survival (PFS) | From baseline to disease progression by Response Evaluation Criteria of Solid Tumors Version 1.1 (RECIST 1.1) or death (up to approximately 2 years)
  PFS is defined as time between the date of first dose of pembrolizumab and the date of either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Overall Survival (OS) | From baseline to approximately 2 years
  OS is defined as time between the date of the first dose of study drug and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shengfa Su, MD,PhD, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, China/Guizhou, China